CLINICAL TRIAL: NCT07072559
Title: Effect of a Dental Simulation Game on Reducing Pain and Anxiety During Primary Teeth Pulpotomy in Pediatric Patients: A Randomized Controlled Clinical Study
Brief Title: Dental Game Impact on Kids' Pulpotomy Pain and Anxiety
Acronym: Electronic
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02012024PP
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pulpotomies Primary Teeth; Anxiety; Pain
Keywords: dental game; pulpotomy; pain; anxiety; tell show do
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Protein-Arginine Deiminases; DC-tell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental simulation game (Experimental): 22 children For the experimental group (group 2) dental simulation game, use the dental simulation game as educational game about procedure this game includes multiple dental procedures like filling cavities, performing root canal treatments, extracting decayed teeth, and conducting orthodontic procedures for animalsAt the first visit children will play on any procedure in dental simulation game, after that the child will be shown two animals, after which they virtually do a root canal procedure. Tasks include performing a dental X-ray, anesthetizing the tooth using a syringe, drilling decayed cavity and start pulp treatment, rinsing, pulp treatment and filling the tooth, applying light cure and finally polishing the teeth . The second visit for pulpotomy procedure will be scheduled two days after first visit. Children will be managed using the TSD (Tell-Show-Do) technique
  Interventions: Other: dental simulation game
- Tell show do (Other): 22 children For the control group (group 1) TSD (Tell-Show-Do) technique group, children will be managed with a verbal explanation and a friendly, non-threatening demonstration of the upcoming dental treatment. The "do" phase involved carrying out the dental procedure as per the prior explanation and demonstration.
  Interventions: Other: tell show do

INTERVENTIONS:
Other: dental simulation game — At the first visit children will play on any procedure in dental simulation game, after that the child will be shown two animals, after which they virtually do a root canal procedure. Tasks include performing a dental X-ray, anesthetizing the tooth using a syringe, drilling decayed cavity and start pulp treatment, rinsing, pulp treatment and filling the tooth, applying light cure and finally polishing the teeth. The second visit for pulpotomy procedure will be scheduled two days after first visit. Children will be managed using the TSD (Tell-Show-Do) technique.
  Other Names: dental game; I pad; electronic device
  Arms: Dental simulation game
Other: tell show do — For the control group (group 1) TSD (Tell-Show-Do) technique group, children will be managed with a verbal explanation and a friendly, non-threatening demonstration of the upcoming dental treatment. The "do" phase involved carrying out the dental procedure as per the prior explanation and demonstration
  Other Names: tell; show; do
  Arms: Tell show do

SUMMARY:
The aim of this study is to evaluate the effect of a dental simulation game on reducing pain and anxiety during primary teeth pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* 1- Children aged between 4 to 7 years of both sexes. 2- Children with behavior rating score 2 and 3 according to Frankl's behavior rating scale.

  3- Children with carious lesions indicated for pulpotomy. 4- Restorable primary lower molars.

Exclusion Criteria:

* 1- Children with special health care needs. 2- Children suffering from systemic diseases.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Frankl's behavior scale | behavior of child will be assessed at baseline .same visit
  The behavior of child will be assessed before treatment, after administration of local anesthesia and finally after pulpotomy using Frankl's behavior rating scale
Venham scale | anxiety of child will be assessed at baseline .same visit
  Anxiety levels of child patient will be assessed by Venham scale. First, explain to patient of all group to select most suitable face that matched with level of anxiety after administration of local anesthesia and after pulpotomy procedure done.
Wong baker scale | pain level of child will be assessed at baseline .same visit
  Pain levels of child patient will be assessed after administration of local anesthesia and finally after pulpotomy using Wong baker scale
pulse rate | vital sign of child will be assessed at baseline.same visit
  Measuring the pulse rate will be by using finger pulse oximeter before treatment, after administration of local anesthesia and at the end of pulpotomy

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of Dentistry, Mansoura University, Al Mansurah, Egypt